CLINICAL TRIAL: NCT03447171
Title: Prospective Evaluation of a Smartphone Application, GoCheckKids™, to Detect Amblyopia Risk Factors in Young Children
Status: Completed | Type: Observational
Sponsor: Gobiquity Mobile Health (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-001
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Amblyopia
Keywords: Amblyopia; Myopia; Hyperopia; Risk Factors; Amblyopia Risk Factors; Smartphone Application (App); Photoscreening; Vision Screening; Mobile Vision Screening; Vision Screening App; Preschool children; Objective vision screening
MeSH Terms: conditions — Amblyopia; Myopia; Hyperopia; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Refractive Error
  Interventions: Device: App Vision Screening

INTERVENTIONS:
Device: App Vision Screening — Using GoCheck Kids App Vision Screening to detect Amblyopia Risk Factors

SUMMARY:
The objective is evaluation of GoCheck Kids, a smartphone application ('App'), for use as a photo screening device in a pediatric population to detect amblyopia risk factors (ARFs).

DETAILED DESCRIPTION:
Detection of amblyopia risk factors using photo screening app in children of ages from 12 months to 8 years

ELIGIBILITY:
Inclusion Criteria:

* Age 12 months to 8 years inclusive.
* Informed consent given by parent or legal guardian.

Exclusion Criteria:

- History of ocular surgery and any condition that would preclude the ability of the investigator to obtain a reliable image and measurement

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study population will be selected from eye clinics.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of amblyopia risk factors detected by Photorefraction | 1 day
  Identification of risk factors compared to gold standard cycloplegic refraction

SECONDARY OUTCOMES:
Number of patients with gaze error identified by photo screening | 1 day
  Detection of gaze error compared to cover test examination results

CONTACTS AND LOCATIONS:
Overall Officials: Sean Donahue, MD, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Alaska Children's Eye & Strabismus, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: Undecided